CLINICAL TRIAL: NCT06192979
Title: Optimize First-line Treatment for Systemic Light Chain Amyloidosis With t (11; 14)
Brief Title: Optimize First-line Treatment for AL Amyloidosis With t (11; 14)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jin Lu, MD (Other)
Responsible Party: Sponsor-Investigator, Jin Lu, MD, Principal Investigator, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023PHB319-001
Record Dates: First submitted 2023-12-12; First posted 2024-01-05 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Amyloidosis; Systemic; AL Amyloidosis
Keywords: t(11;14); Rapid Response; AL amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — daratumumab; Bortezomib; Dexamethasone; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rapid Response Group (Other): Daratumumab, bortezomib, dexamethasone
  Interventions: Drug: Daratumumab; Drug: Bortezomib; Drug: Dexamethasone
- Non-Rapid Response Group (Other): Daratumumab, venetoclax, dexamethasone
  Interventions: Drug: Daratumumab; Drug: Dexamethasone; Drug: Venetoclax

INTERVENTIONS:
Drug: Daratumumab — Daratumumab 16 mg/kg was administered intravenously weekly in cycles one and two, every two weeks for cycles three to six, for at least 6 cycles.
  Daratumumab and hyaluronidase-fihj 1800mg is allowed according to the patients' choice.
Drug: Bortezomib — All patients received 1.0-1.3 mg/m2 subcutaneous bortezomib once weekly of 28 days each for at 6 cycles.
  Arms: Rapid Response Group
Drug: Dexamethasone — All patients received 20-40 mg oral or intravenous dexamethasone
Drug: Venetoclax — All patients received venetoclax 400mg daily.
  Arms: Non-Rapid Response Group

SUMMARY:
Achievement of complete hematologic response (CHR) is vital for systemic AL amyloidosis. Currently, the CHR rate of daratumumab, bortezomib, and dexamethasone (DBD) is close to 60%. Considering that Bcl-2 inhibitor is effective for AL amyloidosis with t(11; 14) and the median hematologic onset time of DBD is 7 days. We design a a prospective study on AL amyloidosis with t(11; 14). All patients receive DBD at the beginning. Patient will receive DBD for at least 6 cycles if achieve rapid hematologic response at day 7, while other patients will receive daratumumab, venetoclax and dexamethasone.

DETAILED DESCRIPTION:
The goal of this clinical trial is to optimize the first line treatment for systemic AL amyloidosis with t(11;14). The aim of this study is to pursue early complete hematologic response. The primary endpoint is overall complete hematologic response (CHR) rate at 6 months. Participants will be treated according to the hematologic response after 7 days. If the patient get rapid response after 7 days, he/she will receive daratumumab, venetoclax and dexamethasone (DBD) for at least 6 cycles. If the patient do not get rapid response, he/she will receive daratumumab, venetoclax and dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of systemic AL amyloidosis;
2. Daratumumab, bortezomib, dexamethasone used in 1st line treatment;
3. Life expectancy greater than 12 weeks;
4. HGB ≥70g/L;
5. Blood oxygen saturation >90%;
6. Total bilirubin (TBil) ≤3×upper limit of normal (ULN); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3.0×ULN;
7. Informed consent explained to, understood by and signed by the patient.

Exclusion Criteria:

1. Fulfill with the criteria of active multiple myeloma or active lymphoplasmacytic lymphoma.
2. Presence of other tumors which is/are in advanced malignant stage and has/have systemic metastasis;
3. Severe or persistent infection that cannot be effectively controlled;
4. Presence of severe autoimmune diseases or immunodeficiency disease;
5. Patients with active hepatitis B or hepatitis C ([HBVDNA+] or [HCVRNA+]);
6. Patients with HIV infection or syphilis infection;
7. Any situations that the researchers believe will increase the risks for the subject or affect the results of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall CHR rate at 6 months | Overall CHR rate at 6 months
  Overall complete hematologic response rate at 6 months

SECONDARY OUTCOMES:
Cardiac response at 6 months | Cardiac response at 6 months
  Cardiac response at 6 months
Renal response at 6 months | Renal response at 6 months
  Renal response at 6 months
Hepatic response at 6 months | Hepatic response at 6 months
  Hepatic response at 6 months
Estimated 2-year PFS | Estimated 2-year PFS
  Estimated 2-year progression free survival
Estimated 2-year OS | Estimated 2-year overall survival
  Estimated 2-year overall survival
MRD status at 6 months | MRD status at 6 months
  Minimal residual disease status at 6 months
TRAEs | TRAEs
  treatment-related adverse events up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jin Lu, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China